CLINICAL TRIAL: NCT00059722
Title: A Phase II, Randomized Double-blind, 2-part, Multicenter Study to Compare the Efficacy of ZD6474 With the Efficacy of ZD1839 (Iressa™) in Subjects With Locally Advanced or Metastatic (IIIB/IV) Non-small Cell Lung Cancer After Failure of First-line Platinum-based Chemotherapy and to Assess the Activity of ZD6474 in Subjects Following Failure of Treatment With ZD1839.
Brief Title: This Study is to Compare the Efficacy of ZD6474 and ZD1839 in Subjects With NSCLC.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6474IL/0003; NCT00072423 (obsolete NCT alias)
Record Dates: First submitted 2003-05-02; First posted 2003-05-05 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; locally advanced or metastatic; second-line
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — vandetanib; Gefitinib

INTERVENTIONS:
Drug: ZD6474
Drug: Placebo
Drug: ZD1839

SUMMARY:
The purpose of this study is to compare the efficacy of ZD6474 and ZD1839 in patients with NSCLC after Failure of Prior Platinum-based Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Failure of either first-line and/or second-line chemotherapy either of which was platinum-based (the prior regimen must have failed the subject because of toxicity or progression of tumor
* Prior histologic or cytologic confirmation of locally advanced or metastatic (IIIB/IV) NSCLC

Exclusion Criteria:

* Subjects who have received second-line or subsequent chemotherapy
* Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic, need not be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2003-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes:
Part A
i. Time to progression
ii. Incidence, CTC grade and type of Aes, clinically significant laboratory abnormalities or changes in vital signs, and ECG changes
Part B

SECONDARY OUTCOMES:
Secondary Outcomes:
Part A
i. Objective response
ii. Disease control at 8 weeks
iii. Time to death
iv. WHO performance status
v. QOL and LCS from the FACT-L questionnaire
Part B
i. Objective response in subjects following treatment with the alternate study treatment
ii. Disease control at 8 weeks in subjects following treatment with the alternate study treatment
iii. WHO performance status in subjects following treatment with the alternate study treatment
iv. QOL and LCS from the FACT-L questionnaire in subjects following treatment with the alternate study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (48):
- United States (18):
  - Research Site, Pine Bluff, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, San Diego, California
  - Research Site, Boca Raton, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Saint Loius, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Madison, Wisconsin
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Mendoza
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Edegem
  - Research Site, Liège
  - Research Site, Wilrijk
- Germany (9):
  - Research Site, Hamburg, Hamburg
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Berlin, State of Berlin
  - Research Site, Ryhope, Sunderland
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Mainz
- South Africa (8):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Lyttelton Manor
  - Research Site, Parktown
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- United Kingdom (5):
  - Research Site, Northwood, Middlesex
  - Research Site, Cardiff, South Glamorgan
  - Research Site, Edinburgh
  - Research Site, Leeds
  - Research Site, Manchester